CLINICAL TRIAL: NCT07174921
Title: Laparoscopic Lateral Suspension Versus Laparoscopic Sacrocolpopexy for Post-Hysterectomy Vaginal Cuff Prolapse: A Randomized Controlled Trial
Brief Title: Post-hysterectomy Vaginal Cuff Prolapse Repair
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ozan Karadeniz, Principal Investigator, Başakşehir Çam & Sakura City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSC Hospital
Record Dates: First submitted 2025-09-07; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Vaginal Cuff Complications
Keywords: prolapse; vaginal cuff; lateral suspension; sacrocolpopexy
MeSH Terms: conditions — Prolapse

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic Sacrocolpopexy (Active Comparator)
  Interventions: Procedure: Laparoscopic Sacrocolpopexy
- Laparoscopic Lateral Suspension (Experimental)
  Interventions: Procedure: Laparoscopic Lateral Suspension

INTERVENTIONS:
Procedure: Laparoscopic Lateral Suspension — Participants in this arm will undergo laparoscopic lateral suspension for post-hysterectomy vaginal cuff prolapse. The procedure involves attaching a synthetic mesh from the vaginal cuff to the lateral abdominal wall to provide support and restore normal vaginal anatomy. Standard perioperative care, including anesthesia and postoperative pain management, will be provided.
  Other Names: Lateral Suspension (Apical Suspension)
  Arms: Laparoscopic Lateral Suspension
Procedure: Laparoscopic Sacrocolpopexy — Participants in this arm will undergo laparoscopic sacrohysteropexy for post-hysterectomy vaginal cuff prolapse. The procedure involves suspending the vaginal cuff to the sacral promontory using a synthetic mesh, restoring vaginal support. Standard perioperative care, including anesthesia and postoperative pain management, will be provided.
  Arms: Laparoscopic Sacrocolpopexy

SUMMARY:
This study is a randomized controlled trial comparing two minimally invasive surgeries-laparoscopic lateral suspension and laparoscopic sacrocolporopexy-for women who develop vaginal cuff prolapse after hysterectomy. Vaginal cuff prolapse occurs when the top of the vagina loses support after the uterus is removed, which can cause discomfort, bulging, or urinary and bowel problems.

The goal of this study is to determine which surgical approach is safer, more effective, and improves quality of life for patients. Women enrolled in the trial will be randomly assigned to one of the two surgeries, and outcomes such as prolapse recurrence, complications, recovery time, and patient satisfaction will be carefully monitored.

By comparing these two techniques, this study aims to provide clear guidance for surgeons and patients to make informed decisions about the best surgical treatment for post-hysterectomy vaginal cuff prolapse.

DETAILED DESCRIPTION:
This study is a randomized controlled trial (RCT) designed to compare the outcomes of two minimally invasive surgical techniques-laparoscopic lateral suspension and laparoscopic sacrocolpopexy-for the treatment of vaginal cuff prolapse following hysterectomy. Vaginal cuff prolapse occurs when the top of the vagina loses its normal support after the uterus has been removed, leading to symptoms such as a sensation of vaginal bulging, pelvic pressure, urinary or bowel dysfunction, and discomfort during daily activities or sexual intercourse.

Eligible participants are women who have previously undergone hysterectomy and are experiencing symptomatic vaginal cuff prolapse. Participants will be randomly assigned to undergo either laparoscopic lateral suspension or laparoscopic sacrocolpopexy. Both procedures are performed using minimally invasive laparoscopic techniques, which typically result in smaller incisions, less pain, and faster recovery compared to traditional open surgery.

The study will assess multiple clinical and patient-reported outcomes, including:

Anatomical success: Prevention of prolapse recurrence at follow-up visits.

Functional outcomes: Improvement in urinary, bowel, and sexual function.

Complications: Intraoperative and postoperative adverse events.

Recovery metrics: Length of hospital stay, return to daily activities, and postoperative pain.

Patient satisfaction: Quality of life and overall satisfaction with the procedure.

By conducting this study, researchers aim to provide evidence-based guidance on which surgical approach offers better long-term outcomes, fewer complications, and higher patient satisfaction. The results of this trial may help clinicians make informed decisions and improve the care of women with post-hysterectomy vaginal cuff prolapse.

ELIGIBILITY:
Inclusion Criteria:

Women aged ≥18 years.

History of hysterectomy (any approach: abdominal, vaginal, or laparoscopic).

Symptomatic vaginal cuff prolapse (POP-Q stage ≥ II).

Able to provide written informed consent.

Willing and able to comply with study procedures and follow-up visits.

Exclusion Criteria:

Prior sacrocolpopexy or lateral suspension surgery.

Active pelvic infection or untreated malignancy.

Severe cardiopulmonary or systemic disease that contraindicates laparoscopic surgery.

Known allergy to mesh materials used in the procedures.

Inability to complete patient-reported questionnaires due to cognitive or language barriers.

Concurrent pelvic organ prolapse requiring additional surgical repair beyond vaginal cuff suspension.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
Anatomical Success (Point C of POP-Q System) | 12 months post-surgery
  Vaginal cuff support measured objectively using POP-Q system, focusing on point C (position of the vaginal apex relative to the hymen). Success is defined as point C remaining above the hymen at follow-up by a blinded examiner.

SECONDARY OUTCOMES:
Operative Time | During surgery
  Total duration of the surgery measured in minutes from incision to closure.
Postoperative Hospital Stay | From the day of surgery through hospital discharge (an expected average of 2 days)
  Length of hospital stay in days from surgery to discharge.
Postoperative Complications | Up to 12 months post-surgery
  Includes mesh exposure, infection, bleeding, urinary or bowel injury, and reoperation.
Pelvic Floor Distress Inventory (PFDI-20) | Preoperative and 12 months post-surgery
  Patient-reported measure of prolapse, urinary, and bowel symptoms.
  The PFDI-20 consists of 3 subscales:
  Pelvic Organ Prolapse Distress Inventory (POPDI-6)
  Colorectal-Anal Distress Inventory (CRADI-8)
  Urinary Distress Inventory (UDI-6) Each subscale is scored 0-100, and the total score is the sum of the three subscales (0-300).
  0 = no pelvic floor-related distress at all.
  300 = the maximum possible distress, meaning the respondent endorsed the highest level of bother on all 20 items.
Pelvic Floor Impact Questionnaire (PFIQ-7) | Preoperative and 12 months post-surgery
  Patient-reported measure of the impact of pelvic floor disorders on daily activities, relationships, and quality of life.
  The PFIQ-7 includes 3 subscales:
  Urinary Impact Questionnaire (UIQ-7)
  Colorectal-Anal Impact Questionnaire (CRAIQ-7)
  Pelvic Organ Prolapse Impact Questionnaire (POPIQ-7)
  Each subscale contains items scored 0-3 ("not at all" to "quite a bit"), then converted to a 0-100 scale.
  The three subscales are summed for a total score ranging from 0 to 300.
  0 = no impact on quality of life.
  300 = maximum impact across all domains (urinary, colorectal-anal, and prolapse).
  Higher scores indicate worse quality-of-life impairment due to pelvic floor disorders.
Patient Global Impression (PGI) Scale | Preoperative and 12 months post-surgery
  Patient-reported scale evaluating overall improvement or satisfaction with surgery, typically rated from 1 ("very much improved") to 7 ("very much worse").

CONTACTS AND LOCATIONS:
Locations (1):
- Basaksehir Cam and Sakura City Hospital, Istanbul, Istanbul, Turkey (Türkiye)